CLINICAL TRIAL: NCT04902846
Title: Application of Biomarkers of Renal Damage in Patients Treated With Immune Checkpoint Inhibitors
Brief Title: Immune Checkpoint Inhibitors Nephrotoxicity
Status: Recruiting | Type: Observational
Sponsor: R. Laura Vicente Vicente (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other); Hospital Clínico Universitario de Valladolid (Other); University of Salamanca (Other)
Responsible Party: Sponsor-Investigator, R. Laura Vicente Vicente, University professor, Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León
Organization: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Other Study IDs: ICITOX
Record Dates: First submitted 2021-05-19; First posted 2021-05-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Kidney Injury; Antineoplastics Toxicity
Keywords: Diagnosis; Nephrotoxicity; Prevention; Oncology; Immune check point inhibitors
MeSH Terms: conditions — Disease; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In this project, only urine samples will be collected. This will be centrifuged, aliquoted and stored at -80 degrees Celsius until its determination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control (no kidney injury): Patients who receive ICI but no develop kidney injury
  Interventions: Diagnostic Test: Early kidney damage biomarkers; Diagnostic Test: Predisposition to kidney injury biomarkers
- Case (kidney injury): Patients who receive ICI and develop kidney injury
  Interventions: Diagnostic Test: Early kidney damage biomarkers; Diagnostic Test: Predisposition to kidney injury biomarkers

INTERVENTIONS:
Diagnostic Test: Early kidney damage biomarkers — In the urine samples of these patients, a series of biomarkers of early kidney damage and / or predisposition to kidney damage will be measured.
  Other Names: albumin; N-acetyl-beta-D-glucosaminidase (NAG); Kidney Injury Molecule-1 (KIM-1); Neutrophil gelatinase-associated lipocalin (NGAL)
Diagnostic Test: Predisposition to kidney injury biomarkers — In the urine samples of these patients, a series of biomarkers of predisposition to kidney damage will be measured.
  Other Names: Transferrin; Ganglioside GM2 activator isoform 1 (GM2AP)

SUMMARY:
In recent years, immunotherapy has been postulated as one of the most effective strategy in the fight against cancer. The greatest success in this field has been achieved through the inhibition of molecules involved in the brake of the adaptive immune response. The compounds capable of blocking the action of these molecules constitute the "immune checkpoint inhibitors" (ICI). Despite its efficacy, the treatment with ICI causes adverse effects, and in the case of kidney damage, the prognosis has been shown to worsen in cancer patients who develop renal dysfunction. Currently, the diagnosis based on laboratory tests is insufficient to predict the underlying kidney injury and identify the type of damage. The hypothesis proposed that the renal lesion could be subclinical, and therefore the possibility of using new urinary biomarkers could be a useful diagnostic tool that would allow these patients to be managed in a preventive (risk markers) and early way (early markers), and even to elucidate if renal damage is due to this therapy or to other factors (differential diagnostic markers). To develop this hypothesis it is proposed to validate biomarkers in patients treated with ICI by developing a prospective study. The diagnostic products derived from this study will improve the clinical practice of cancer treatment with ICI, and therefore the expectancy and quality of life of patients.

DETAILED DESCRIPTION:
During the last decade, advances in the knowledge of both the immune response to tumors, as well as the understanding of their evasion mechanisms, has made it possible to design treatments aimed at improving said response and increasing patient survival in figures up to now unthinkable. The greatest success in this field has been achieved through the inhibition of molecules involved in the braking of the adaptive immune response: the so-called CTLA-4 (cytotoxic T-lymphocyte antigen-4) and PD-1 (programmed cell death protein-1), with their respective ligands. The compounds capable of blocking the action of these molecules constitute the so-called "immune checkpoint inhibitors" (ICI).

As with conventional therapies, the adverse effects that these drugs develop in many cases limit their use. Although nephrotoxicity is less common than other complications (liver, gastrointestinal, skin, and lung toxicity), kidney effects have been shown to worsen prognosis in cancer patients who develop kidney dysfunction. In addition, therapies based on ICI combinations have recently been promoted to avoid the resistance acquired by the tumor to treatment, and have even been associated with chemotherapy, which has improved the response, but has increased the risk of nephrotoxic adverse events.

Kidney injury due to immunotherapy treatment is characterized by acute kidney damage, proteinuria, electrolyte disturbances, tubular injuries, glomerular injuries, and more frequently acute tubulointerstitial nephritis, the toxic mechanisms underlying these events are largely unknown. The usual clinical procedure when kidney damage appears is to suspend immunotherapy treatment and administer systemic corticosteroids. However, discontinuation of treatment may not be appropriate without diagnostic confirmation of the progression of kidney damage, but continuation of treatment if the diagnosis is subsequently confirmed may lead to definitive and irreversible kidney damage.

At present, the diagnosis of kidney injury based on clinical findings and laboratory tests is insufficient to predict the underlying kidney injury and identify the type of damage, since serum markers such as creatinine or urea only provide information when the damage is already established. In addition, it must be taken into account that kidney injuries, such as ischemic and / or nephrotoxic tubular injury, paraneoplastic kidney injury, glomerular injuries, and tubular obstruction can occur in cancer patients as a consequence of their pathology and associated therapy. . Therefore, a careful evaluation of the possible causes should be made to make the correct diagnosis in patients undergoing treatment with ICI (for example, interstitial nephritis due to ICI versus other types of damage by other drugs) and based on that, proceed to the management of the patient optimally. In this scenario, renal biopsy is presented as the only alternative to definitively diagnose the lesion and potentially guide therapy. Although it is the definitive diagnostic method, it is an invasive technique, not without complications, therefore the possibility of using biomarkers capable of identifying the type of damage (differential diagnosis biomarkers) would represent a highly relevant diagnostic advance.

Another important approach in diagnosis is the identification of damage early, since creatinine levels (a commonly used marker) do not show a significant increase until kidney function has already decreased by 50%. Currently, the usefulness of biomarkers of early kidney damage associated with drug treatment has been described. These markers are components or metabolic derivatives, degradation compounds or remains of them that appear in the urine as a consequence of damage to kidney structures, showing subclinical damage.

A significant advance in the management of kidney injury would be to find markers capable of identifying subjects at risk, that is, in a stage prior to damage (risk biomarkers). It has been defined that different drugs and kidney toxins, in completely subtoxic doses, are capable of predisposing, or making experimental animals more sensitive to acute kidney damage. The relevance of this situation is that individuals apparently unaffected by the adverse effects of a treatment, or by exposure to a substance, could be, without knowing it and therefore unable to do anything to prevent it, exposed to developing kidney damage acute in situations, or under certain circumstances (other treatments, radiological contrasts, environmental toxins, etc.) that do not produce any harm in non-predisposed individuals. Associated with this condition, it have been identified and patented, and are clinically and technologically developing urinary markers related to this acquired hypersensitivity. Their clinical application would allow, not only to detect this predisposition, but also to stratify patients in a preventive and personalized way, according to the individual risk they acquire as a consequence of apparently innocuous pharmacological treatments or other circumstances inherent to their pathology. On this basis, it is proposed in this project to explore possible biomarkers that can be detected by patients at risk before starting treatment with ICI.

For all the above, this project will be carried out through preclinical and clinical studies. The main objective proposed in clinical setting is to validate biomarkers as diagnostic tools for kidney damage in patients treated with immune checkpoint inhibitors:

1.1. Before starting treatment to detect patients at risk (risk markers) 1.2. During treatment, in a first phase to detect early lesions (early biomarkers)

With this objective, it is intended to study whether these biomarkers can be a valid tool in the management of kidney damage in patients treated with ICI, responding to an unresolved diagnostic need.

PATIENT DATA COLLECTION

A database will be prepared that collects the following variables for each patient: age, sex, family history, personal history, tumor type, antitumor treatment regimen, clinical characteristics of the case, comorbidity factors, allergies, usual medication, occasional drugs and follow-up data.

Urine Sampling

The study times, in which urine samples will be taken, will be as follows:

* Before each antineoplastic cycle (Pre ICI)
* One week after each antineoplastic cycle (Post ICI)

Processing and storage of urine samples In the case of samples from the Salamanca University Hospital, the samples will be handled and kept in the Sample Bank of the Salamanca University Clinical Hospital. The samples from the Valladolid University Clinical Hospital will be handled and kept in the Oncology Service itself. After collection, the samples will be centrifuged to remove possible sediments and later frozen in several aliquots at -80 degrees Celsius.

Study of kidney function using clinical parameters At all times of the study, the plasma concentration of creatinine, urea and electrolytes will be extracted from the analytics issued by the Biochemistry Service of the respective hospitals. These tests are prescribed by doctors as part of the patient care process.

Study of early markers and risk markers of acute kidney damage The rest of the analytical determinations necessary for the study will be carried out in the laboratory of the "Theranostic Unit of Renal and Cardiovascular Diseases" of IBSAL. They are the following: urinary creatinine concentration (commercial kit), creatinine clearance (using conventional mathematical formulas), proteinuria, (Bradford technique), urinary NAG excretion (using colorimetric kit), KIM-1, NGAL, albumin, transferrin and GM2AP (by ELISA or Western blot).

STATISTICAL ANALYSIS Data analysis will be done with "SPSS 25.0". A significance level of 0.05 will be used. Different contrasts will be applied depending on the association to be studied in each case, and the type of variables, such as: normality test (Kolmogorov-Smirnov, Shapiro-Wilk), frequency comparison (χ2), correlation test (Pearson, Spearman), comparison of means for independent data (ANOVA and Kruskal-Wallis) and ANOVA for repeated measures and Wilcoxon test for paired data. Finally, to simultaneously study data sets with several variables measured for each individual or parameter collected, techniques with Multivariate Analysis will be used, such as: regression analysis, general linear models, binary logistic regression and correspondence analysis.

STUDY LIMITATIONS The variables included are biomarkers of early kidney damage and of predisposition to acute kidney damage induced by certain kidney toxins. It is possible that there are other (unknown) markers, not analyzed, and which can predict, diagnose earlier or allow a differential etiological diagnosis of kidney damage associated with treatment with immunotherapy or immunotherapy / chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients waiting for immunotherapy or combination immunotherapy / platinum compounds

Exclusion Criteria:

* Patients who are terminally ill
* Patients who do not wish to sign the informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will receive ICI as part of a diagnostic or interventional procedure
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2021-05-19 (Actual); Primary Completion 2028-04-23 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of urinary albumin | During 1 year at the times: pre ICI (before administering each cycle of ICI) and post ICI (one week after each administration of ICI)
  It is a biomarker of early kidney damage. It is able to detect kidney damage in the early stages, before the clinical markers creatinine and plasma urea. There are no reference values for humans, so the means of non-smoking patients without risk factors (group 1) should be compared with the rest of the groups. This biomarker will be measured at different times to evaluate its evolution and compare it against the baseline value.
Change of urinary N-Acetyl-β-D-Glucosaminidase (NAG) | During 1 year at the times: pre ICI (before administering each cycle of ICI) and post ICI (one week after each administration of ICI)
  It is an enzyme whose urinary excretion is elevated in case of kidney damage. It is capable of detecting damage before the classic plasma creatinin and urea markers. There are no reference values for humans, so the means of non-smoking patients without risk factors (group 1) should be compared with the rest of the groups. This biomarker will be measured at different times to evaluate its evolution and compare it against the baseline value.
Change of urinary Kidney Injury Molecule-1 (KIM-1) | During 1 year at the times: pre ICI (before administering each cycle of ICI) and post ICI (one week after each administration of ICI)
  It is a biomarker of early kidney damage. It is able to detect kidney damage in the early stages, before the clinical markers creatinine and plasma urea. There are no reference values for humans, so the means of non-smoking patients without risk factors (group 1) should be compared with the rest of the groups. This biomarker will be measured at different times to evaluate its evolution and compare it against the baseline value.
Change of urinary Neutrophil gelatinase-associated lipocalin (NGAL) | During 1 year at the times: pre ICI (before administering each cycle of ICI) and post ICI (one week after each administration of ICI)
  It is a biomarker of early kidney damage. It is able to detect kidney damage in the early stages, before the clinical markers creatinine and plasma urea. There are no reference values for humans, so the means of non-smoking patients without risk factors (group 1) should be compared with the rest of the groups. This biomarker will be measured at different times to evaluate its evolution and compare it against the baseline value.
Change of urinary biomarkers of predisposition to kidney injury | During 1 year at the times: pre ICI (before administering each cycle of ICI) and post ICI (one week after each administration of ICI)
  It is a group of markers that are in patent phase so their names can not be mentioned. They are able to detect the susceptibility to kidney damage before administering a nephrotoxic agent. There are no reference values for humans, so the means of non-smoking patients without risk factors (group 1) should be compared with the rest of the groups. This biomarker will be measured at different times to evaluate its evolution and compare it against the baseline value.

SECONDARY OUTCOMES:
Body weight | These data will be collected once, at time 0 (moment of enrollment in the study)
  Body weight will be measured to each patient and expressed in kilograms
Height | These data will be collected once, at time 0 (moment of enrollment in the study)
  The height will be measured to each patient and expressed in meters
Body mass index (BMI) | These data will be collected once, at time 0 (moment of enrollment in the study)
  Weight and height will be combined to report BMI in kg/m^2
Age | These data will be collected once, at time 0 (moment of enrollment in the study)
  Through the year of birth, the patient's age will be calculated, which will be expressed in years.
Gender | These data will be collected once, at time 0 (moment of enrollment in the study)
  Patients will be classified in Male or Female
Concentration of plasma creatinine | These data will be collected once, at time 0 (moment of enrollment in the study)
  From the analytical biochemistry performed on the patient as part of his usual procedure, the plasma urea data will be obtained in mg/dL units.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Isabel Morales Martín, PhD, Principal Investigator — University of Salamanca
Locations (2):
- Spain (2):
  - Servicio de Oncología del CAUSA, Salamanca
  - Servicio de oncología del Hospital Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vicente-Vicente L, Casanova AG, Tascon J, Prieto M, Morales AI. New Challenges in the Diagnosis of Kidney Damage Due to Immune Checkpoint Inhibitors Therapy: An Observational Clinical Study. Diagnostics (Basel). 2023 Jul 28;13(15):2524. doi: 10.3390/diagnostics13152524. PMID 37568887

DOCUMENTS (1):
  • Informed Consent Form (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/46/NCT04902846/ICF_000.pdf